CLINICAL TRIAL: NCT06283186
Title: Differences in Exercise-Induced Hypoalgesia at Local and Distal Levels Using Lower and Upper Limb Cycle Ergometer Protocols: A Randomized Controlled Trial in Healthy Participants
Brief Title: Comparative Exercise-Induced Hypoalgesia in Upper and Lower Limbs: A Randomized Controlled Trial in Healthy Individuals
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Centro Universitario La Salle (Other)
Responsible Party: Principal Investigator, Álvaro Reina Varona, Principal Investigator, Centro Universitario La Salle
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSEULS-PI-004/2024
Record Dates: First submitted 2024-02-22; First posted 2024-02-28 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Healthy Subjects
Keywords: Local Hypoalgesia; Distal Hypoalgesia; Aerobic Exercise; Pressure Pain Thresholds
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lower limb cycle ergometer (Experimental): The participants in the lower limb cycle ergometer group will undergo a 30-minute aerobic exercise intervention comprising a 5-minute warm-up, 20 minutes of training at 70-80% of the heart rate reserve, and a 5-minute cool-down.
  Interventions: Other: Aerobic exercise
- Upper limb cycle ergometer (Experimental): The participants in the upper limb cycle ergometer group will undergo a 30-minute aerobic exercise intervention comprising a 5-minute warm-up, 20 minutes of training at 70-80% of the heart rate reserve, and a 5-minute cool-down.
  Interventions: Other: Aerobic exercise
- Control (No Intervention): Participants in the control group will remain seated for the entire 30-minute duration of the experiment without receiving any form of distraction.

INTERVENTIONS:
Other: Aerobic exercise — Aerobic exercise with lower limb cycle ergometer
  Arms: Lower limb cycle ergometer
Other: Aerobic exercise — Aerobic exercise with upper limb cycle ergometer
  Arms: Upper limb cycle ergometer

SUMMARY:
This randomized controlled trial with healthy subjects aims to compare exercise-induced hypoalgesia among three groups: one utilizing a lower limb cycle ergometer, another using an upper limb cycle ergometer, and a control group. The exercise protocol involves 30 minutes of aerobic activity at 70-80% of the heart rate reserve. Exercise-induced hypoalgesia will be assessed by measuring pressure pain thresholds in the thigh and elbow. Additionally, a secondary objective is to compare the lower limb and upper limb cycle ergometer groups in terms of their effects on pressure pain thresholds in the thigh and elbow. Thus, the study anticipates observing differences in local and distal hypoalgesia based on the trained region.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic subjects aged between 18 and 64 years.

Exclusion Criteria:

* Cardiovascular, respiratory, metabolic, neurological, or osteomuscular signs or pathologies.
* History of epilepsy.
* Pregnant
* Pharmacological treatment.
* Participants who present any type of pain on the day of the measurements or who have frequently suffered pain during the previous 12 weeks.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Pressure pain threshold (PPT) on dominant quadriceps and dominant lateral epicondyle | Three measurementes: before, immediately after intervention, and 30 minutes after intervention
  PPT is tested on the muscle belly of the quadriceps on the dominant side, 10 centimeters cranial to the superior pole of the patella, and on the muscle belly of the epicondyle muscles on the dominant side, 5 centimeters caudal to the epicondyle. The region to be pressed is marked with a pen. The patient is instructed to report the first appearance of the sensation of "discomfort". An ascending ramp of 0.5 kg/cm/s is applied, at the rhythm of a metronome. The measurement is started on the quadriceps and alternated with the epicondyle until 3 measurements of each region are obtained. Each measurement in the same region is obtained after 30 seconds of rest. This protocol has demonstrated high inter-observer reliability measuring healthy subjects (ICC = 0.91).

SECONDARY OUTCOMES:
International Physical Activity Questionnaire (IPAQ) | Before intervention (up 5 minutes)
  7-item questionnaire on the level of physical activity at different intensities (high, moderate, and low) and hours sitting. A higher score means higher weekly physical activity.
Fatigue Assessment Scale (FAS) | Before intervention (up 5 minutes)
  10-item questionnaire that allows for the evaluation of the participant's current level of fatigue. A higher score means higher fatigue.
Heart rate | During intervention (up 30 minutes)
  Heart rate will be measured during the procedure by a Polar H10 sensor and a Polar Ignate WR 30M watch.
Rate of perceived exertion (RPE) | Immediately after intervention (up 10 seconds)
  RPE Borg CR-10 is used to measure how hard your body works during physical activity. It runs from 0 - 10, using numbers to rate how much effort an activity takes.
Physical Activity Readiness Questionnaire (PAR-Q) | Before intervention (up 5 minutes)
  7-item questionnaire that assesses an individual's readiness to engage in physical activity based on whether any known contraindications have been ruled out by the participant. If all the questions are negative, the participant can safely engage in a physical activity.

CONTACTS AND LOCATIONS:
Locations (1):
- CSEU LaSalle, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No